CLINICAL TRIAL: NCT03937336
Title: A School-based Randomized Controlled Trial to Promote Cycling to School and Physical Activity in Adolescents: The PACO RCT Study
Brief Title: The PACO RCT Study
Acronym: PACO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); University of Jaén (Other); University of Valencia (Other); University of Castilla-La Mancha (Other); Pontificia Universidad Catolica de Valparaiso (Other); University of Otago (Other)
Responsible Party: Principal Investigator, Palma Chillón Garzón, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DEP2016-75598-R
Record Dates: First submitted 2019-04-10; First posted 2019-05-03 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Physical Activity; Sedentary Lifestyle; Behavior
Keywords: Active Commuting; Health behaviour; Design; School-based intervention; Children; Youth; Self-Determination Theory; Walking
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: Randomized Control Trials
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Bike Intervention Group (Experimental): A 1-month bike-based program (1 session/week)
  Interventions: Behavioral: Bike Intervention Group

INTERVENTIONS:
Behavioral: Bike Intervention Group — A 1-month biking-based program. The biking program consists of 4 sessions/month of 120 min at physical education lessons in school, and will focus on promote biking through theory and practice lessons about cycle training skills including on-road training
  Arms: Bike Intervention Group

SUMMARY:
The aim of this school-based cycling intervention called "Cycling and Walk to School" (PACO, for its Spanish acronym) will be to examine their effects on adolescent's cycling to and from school and physical activity (PA). This study will also examine the effects of this intervention in several active commuting to and from school (ACS)-related variables belonging to Self-Determination Theory (SDT) and Social-Ecological Model (SEM).

DETAILED DESCRIPTION:
This study will also examine the effects of this intervention in several active commuting to and from school (ACS)-related variables belonging to SDT and SEM. In this randomized controlled trial will participate 360 adolescents, belonging to six secondary schools (three experimental and three control) from three Spanish cities. The intervention will be conducted by both the research staff and the physical education (PE) teacher through four cycling sessions (one per week). PA levels will be measured by accelerometers, and the other study variables by using self-reported scales, before and after the intervention programme. The primary outcomes will be: cycling to school, ACS, and PA levels. The secondary outcomes will be: SDT (Self-Determination Theory) -related variables in ACS and individual, interpersonal, communittal and environmental variables related to ACS belonging to SEM (Social-Ecological Model). The findings of this study will provide a comprehensive understanding of the effects of this short-term school-based intervention on cycling to school and PA levels of Spanish adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Have at least one group of 3º ESO with a minimum of 15 students.
2. Obtain a minimum of 15 informed consent to carry out the project in the school.
3. That the students of 3rd ESO had not participated in other interventions in the center on active commuting during the ESO stage.
4. Not having public school transport for students; in this case, the project can not be carried out.

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change of the self-reported Mode of commuting | 1 week during both measurement points (baseline and Post-evaluation)
  Assessment of the mode of commuting using "Mode and Frequency of Commuting To and From School Questionnaire".
Change of the objective Mode of commuting | 1 week during both measurement points (baseline and Post-evaluation)
  Assessment of the mode of commuting using GPS.
Change of the objective Mode of commuting | 1 week during both measurement points (baseline and Post-evaluation)
  Assessment of the mode of commuting using accelerometers.
Change in physical activity levels | 1 week during both measurement points (baseline and Post-evaluation)
  Assessment of physical activity levels using accelerometers.
Change in self-reported physical activity levels | 1 week during both measurement points (baseline and Post-evaluation)
  Assessment of physical activity levels using YAP questionnaire.

SECONDARY OUTCOMES:
Change in Children´s behaviours | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of mode of commuting to/from school using Mode and Frequency of Commuting To and From School Questionnaire. Scale range: active, passive or mix.
Change in Children´s behaviours | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of sleep duration using UP and DOWN Study questionnaire.
Change in Children´s behaviours | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of breakfast consumption using ENERGY Spanish questionnaire and enKids study. Scale range: Healthy or Not Healthy (subscale: yes/no, sum of groups of aliment).
Change in Children´s behaviours | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of accompaniment to school using the question extracted of Herrador-Colmenero et al, 2017.
Change in Children´s behaviours | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of individual factors of Social-Ecological model (Sociodemographics; health status; psychosocial; perception; behaviour) using motivation and behaviour change techniques (MBCTs) used in Self Determination Theory -based interventions (Teixeira et al., 2020).
Change in Children´s behaviours | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of interpersonal factors of Social-Ecological model (Parent's Sociodemography, perception and behaviour; Peer social support; Family SES) using motivation and behaviour change techniques (MBCTs) used in Self Determination Theory -based interventions (Teixeira et al., 2020).
Change in Children´s behaviours | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of community factors of Social-Ecological model (School characteristics; city characteristics) using motivation and behaviour change techniques (MBCTs) used in Self Determination Theory -based interventions (Teixeira et al., 2020).
Change in Children´s behaviours | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of environment factors of Social-Ecological model (Route home-school; home neighbourhood; distance home-school; school neighbourhood) using motivation and behaviour change techniques (MBCTs) used in Self Determination Theory -based interventions (Teixeira et al., 2020).
Change in Children´s perceptions | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of perceived environment using ALPHA environmental ((Instruments for Assessing Levels of PHysical Activity and Fitness) questionnaire. Score is extracted of average of differents items include in the questionnaire.
Change in Children´s perceptions | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of barriers to active commuting to/from school using BATACE(BArreras en el Transporte Activo al Centro Educativo) questionnaire. Score is extracted of average of items include in the questionnaire.
Change in children's psychosocial variables | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of autonomy using BPNES questionnaire (Basic Psychological Needs in Exercise Scale) subscales 1-5. Score is extracted of average of questionnaire.
Change in children's psychosocial variables | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of motivation using BREQ questionnaire (Behavioural Regulation in Exercise Questionnaire) subscales 0 - 4. Score is extracted of average of questionnaire.
Change in children's psychosocial variables | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of relatedness and competence to active commuting to school BPNES questionnaire (Basic Psychological Needs in Exercise Scale) subscales 1-5. Score is extracted of average of questionnaire.
Change in anthropometry | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of height and weight, (e.g., weight and height will be combined to report BMI in kg/m^2).
Change in anthropometry | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of waist circumference in centimetres.
Change in anthropometry | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of neck circumference in centimetres.
Change in parent´s behaviours | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of parent's physical activity using IPAQ (International Physical Activity Questionnaire) short form. Score is extracted of sum of time of physical activity.
Change in parent´s behaviours | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of parent's mode of commuting to work using SRTS (Safe Route to School) questionnaire. Score scale is Active, Pasive or Mix.
Change in parent´s perceptions | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of barriers to active commuting to/from school of their children using PABACS (parental perception of barriers towards active commuting to school) questionnaire. Score is extracted of average of items. Subscale is 0 - 4.
Change in parent´s perceptions | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of perceived environment using ALPHA environmental(Instruments for Assessing Levels of PHysical Activity and Fitness) questionnaire. Score is extracted of average of different items include in the questionnaire.
Change in parent´s perceptions | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of children´s distance to allow them to active commute to/from school using Family questionnaire. Score range is between none - >5km.
Change in parent´s perceptions | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of children´s age to allow them to active commute to/from school using Family questionnaire. Score range is between <7y - >18y.
Change in parent´s perceptions | 1 day during both measurement points (baseline and Post-evaluation)
  Assessment of social support using Family questionnaire. Score range is: none; few; many; everyone.

CONTACTS AND LOCATIONS:
Locations (1):
- Palma Chillón Garzón, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Herrador-Colmenero M, Perez-Garcia M, Ruiz JR, Chillon P. Assessing modes and frequency of commuting to school in youngsters: a systematic review. Pediatr Exerc Sci. 2014 Aug;26(3):291-341. doi: 10.1123/pes.2013-0120. Epub 2014 Apr 10. PMID 24722834